CLINICAL TRIAL: NCT03337893
Title: Investigation of Breastfeeding Protection Against Infant Infections and Childhood Diseases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yildiz Atadag (Other Government)
Responsible Party: Sponsor-Investigator, Yildiz Atadag, Medical Doctor, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: 307
Record Dates: First submitted 2017-10-23; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Breast Feeding; Disease
MeSH Terms: conditions — Breast Feeding; Disease | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breastfed: The kids who breastfed
  Interventions: Diagnostic Test: blood pressure
- non-breastfed: The kids who did not breastfed
  Interventions: Diagnostic Test: blood pressure

INTERVENTIONS:
Diagnostic Test: blood pressure — it will be done both right and left arms

SUMMARY:
Objective: It is widely accepted that breastfeeding (AS) is superior to other forms of nutrition in the first six months of life. Breastmilk contains nutrient items in appropriate quantities and a high bioavailability according to the needs of each baby. The United Nations Children's Fund (UNICEF) and the World Health Organization (WHO) recommend that babies take AS alone and then continue to feed on AS with up to two years of age, with appropriate supplementary nutrition, during the first six months of life.

Even in the hottest climates, breastfeeding babies have been shown to have no additional nutrient or fluid requirements for the first six months, including water. In the first 6 months of breastfeeding with breast milk alone (YAS), the incidence of many diseases, especially infectious diseases, decreases and the brain development is better.

Despite its numerous benefits, mother milk is not utilized in our country sufficiently. According to the Turkish Demographic and Health Survey (TNSA), the rate of breastfeeding in Turkey was 91.8% in Turkey, while the proportion of babies fed only breast milk in the first 6 months was 30.1%.

Infants related deaths, otitis media, lower respiratory tract infections, gastroenteritis, obesity were more common in children who were fed formula milk compared to children who were fed breast milk during the first year of life. Obesity can reduce insulin resistance and hypertension risks later in life.

According to the research done by Kramer and his colleagues on 13889 children, no effect of breastfeeding on physical development, obesity and hypertension was found.

In this study, whether breast feeding was associated with otitis media in the first year, lower respiratory tract infection, gastroenteritis; in the first 5 years of age, obesity and hypertension.

DETAILED DESCRIPTION:
Method: This descriptive study will be conducted by Gaziantep Şahinbey Bağlarbaşı ASM, a 5-year-old children who applied between 01.10.2017 - 04.04.2018, with their weight and blood pressure measurements and their parents' questionnaires. Approximately 500 children will be taken to work. Informed consent is obtained from the parents of the patients who will be employed, and verbal consent is given from the children. Those who do not give their approval will not be included in the study. People with a known congenital disease, those with no birth week between 38 and 42 and a birth weight between 2500 and 4000 grams will not be included in the study.

The length measurement shall be made on a fixed scale, with the back of the head on a flat surface, with the head perpendicular, and with the eyes vertically facing (Frankfurt plane), the distance between the top of the head and the soles of the feet shall be a fixed scale or gauge. Blood pressure measurement will be measured by a digital blood pressure meter from the left and right hand (M6; Omron Healthcare).

Measurements of height, weight and hemoglobin in the past ages of the subjects taken in the study group will be taken from the computer programs used in the family medicine system. Percentile values of measurements belonging to each age group will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being at the age of 5
* birth weight between 2500 and 4000 grams
* birth week is between 38-42 weeks

Exclusion Criteria:

* Not being at the age of 5
* birth week is not between 38-42 weeks
* birth weight between 2500 and 4000 grams
* having a serious illness e.g. cerebral palsy

Ages: 5 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: 5 year old kids
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
BP | Baseline for age 5
  Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Sahinbey Baglarbasi Family Health Center, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Background] Gökçay G, Garipağaoğlu M. Çocukluk ve Ergenlik Döneminde Beslenme. İstanbul: Saga Yayınları, 2002: 24-63.
- [Background] Gökçay G, Garibağaoğlu M. Sağlıklı Çocuğun Beslenmesi. İçinde: Neyzi O, Ertuğrul T: Pediatri. 1. Cilt. İstanbul: Nobel Tıp Kitabevi, 2002: 183-202.
- [Background] American Academy of Pediatrics. Nutrition and Immunitiy. Chapter 31. In: Pediatric Nutriton Handbook CD- ROM. 4 th ed. Elk Growe Village: Abbott Laboratories, 1998: 473-84.
- [Background] Lawrens RA, Lawrence RM. Host-resistance factors and immunologic significance of human milk. In: Lawrens RA, Lawrence RM (eds). Breastfeeding. St. Louis: Mosby, 1994: 159-95.
- [Background] T.C. Sağlık Bakanlığı, Hacettepe Üniversitesi Nüfus Etüdleri Enstitüsü. Türkiye Nüfus ve Sağlık Araştırması 2003. Ankara: Macro International Inc, 2003.
- [Background] Hacettepe Üniversitesi Nüfus Etütleri Enstitüsü (2014), "2013 Türkiye Nüfus ve Sağlık Araştırması". Hacettepe Üniversitesi Nüfus Etütleri Enstitüsü, T.C. Kalkınma Bakanlığı ve TÜBİTAK, Ankara, Türkiye
- [Background] Stuebe A. The risks of not breastfeeding for mothers and infants. Rev Obstet Gynecol. 2009 Fall;2(4):222-31. PMID 20111658
- [Background] Kramer MS, Matush L, Vanilovich I, Platt RW, Bogdanovich N, Sevkovskaya Z, Dzikovich I, Shishko G, Collet JP, Martin RM, Davey Smith G, Gillman MW, Chalmers B, Hodnett E, Shapiro S; PROBIT Study Group. Effects of prolonged and exclusive breastfeeding on child height, weight, adiposity, and blood pressure at age 6.5 y: evidence from a large randomized trial. Am J Clin Nutr. 2007 Dec;86(6):1717-21. doi: 10.1093/ajcn/86.5.1717. PMID 18065591
- [Background] Mazıcıoğlu MM.Büyüme gelişme izleminde kullanılan antropometrik ölçüm yöntemleri: Büyüme takibinin metodolojisi.Türkiye Aile Hekimliği Dergisi 2011;15(3):101-108.
- [Background] Altunkan S, Ilman N, Kayaturk N, Altunkan E. Validation of the Omron M6 (HEM-7001-E) upper-arm blood pressure measuring device according to the International Protocol in adults and obese adults. Blood Press Monit. 2007 Aug;12(4):219-25. doi: 10.1097/MBP.0b013e3280f813d0. PMID 17625394
- [Background] Coleman A, Freeman P, Steel S, Shennan A. Validation of the Omron 705IT (HEM-759-E) oscillometric blood pressure monitoring device according to the British Hypertension Society protocol. Blood Press Monit. 2006 Feb;11(1):27-32. doi: 10.1097/01.mbp.0000189788.05736.5f. PMID 16410738
- [Background] Topouchian JA, El Assaad MA, Orobinskaia LV, El Feghali RN, Asmar RG. Validation of two automatic devices for self-measurement of blood pressure according to the International Protocol of the European Society of Hypertension: the Omron M6 (HEM-7001-E) and the Omron R7 (HEM 637-IT). Blood Press Monit. 2006 Jun;11(3):165-71. doi: 10.1097/01.mbp.0000209078.17246.34. PMID 16702826
- [Background] World Health Organization, UNICEF. Global Strategy for Infant and Young Child Feeding, Geneva: WHO, 2003: 1-4, 7-9.